CLINICAL TRIAL: NCT02277470
Title: Study of the Pharmacokinetics of Golimumab in Moderate to Severe Ulcerative Colitis
Acronym: GO-KINETIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, Hanke Brandse, drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL48785.018.14
Record Dates: First submitted 2014-10-17; First posted 2014-10-29 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Ulcerative Colitis
Keywords: pharmacokinetics, Golimumab, IBD
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples and blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Golimumab: Patients who are eligible for golimumab therapy.

SUMMARY:
The purpose of this study is to gain insights in the pharmacokinetics of golimumab in moderate to severe Ulcerative Colitis after subcutaneous administration, during induction and maintenance treatment the investigators will collect blood and stool samples at different time points.

DETAILED DESCRIPTION:
The pharmacokinetic characteristics of golimumab will be assessed by using blood and stool samples; collected during induction and maintenance treatment Patients will undergo 13-16 blood sample collections, 13-16 stool sample collections and 3 endoscopies during 16 hospital visits in 1 year. They are also asked to fill in a short questionnaire (9x). At endoscopy visits a questionnaire regarding quality of life will be taken.The population pharmacokinetics of golimumab will be assessed using nonlinear mixed-effects modelling (NON-MEM).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years, either male or female
* Moderate to severe UC (according to Mayo score (2 or 3) baseline endoscopy), both anti-TNF naïve and anti-TNF exposed patients will be included
* Baseline endoscopy
* Obtained written informed consent

Exclusion Criteria:

* Contra-indication to golimumab: TBC, severe infections or congestive heart failure.
* Imminent need for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for inclusion are patients (either outpatient or hospitalized) with moderate to severe UC refractory to corticosteroids and immunomodulators.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Golimumab concentrations (peak/trough,AUC) | day 0,1,4,7,14,18, week 4,6,10,18,30,42,52
  By measuring golimumab concentrations at different time point during induction and maintenance therapy we can determine pharmacokinetic parameters of golimumab in ulcerative colitis patients.

SECONDARY OUTCOMES:
Development of Golimumab-antibodies | day 0,1,4,7,14,18, week 4,6,10,18,30,42,52
  Assessment of neutralizing antidrug-antibodies by radiomimmuno assay
Endoscopic response | week 10, 52
  defined by improvement in endoscopic Mayo score of at least 1 point
Clinical response by SCCAI | week 10, 52
Quality of Life by IBDQ, SF-36 | week 10, 52
fecal calprotectin | day 0,1,4,7,14,18, week 4,6,10,18,30,42,52
fecal golimumab levels | day 1,4,7,14,18, week 4,6,8,18,30,42,52
serum CRP | day 0,1,4,7,14,18, week 4,6,10,18,30,42,52
Clearance | day 1,4,7,14,18, week 4,6,10,18,30,42,52
  calculated from primary outcome (concentrations)
serum Albumin | day 0,1,4,7,14,18, week 4,6,10,18,30,42,52

CONTACTS AND LOCATIONS:
Overall Officials: Geert R D'Haens, MD, Phd, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); mark lowenberg, MD, Phd, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Ron Mathot, Phd, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland